CLINICAL TRIAL: NCT04109261
Title: Retrospective Observational Analysis of Palbociclib Treatment in Patients With Advanced Breast Cancer Within a Compassionate Use Programme
Brief Title: Analysis of Palbociclib Treatment in Patients With Advanced Breast Cancer Within a Compassionate Use Programe
Acronym: PALBOCOMP
Status: Completed | Type: Observational
Sponsor: Fernando Moreno Antón (Other)
Responsible Party: Sponsor-Investigator, Fernando Moreno Antón, Principal Investigator, Hospital San Carlos, Madrid
Organization: Hospital San Carlos, Madrid (Other)
Other Study IDs: PALBOCOMP
Record Dates: First submitted 2019-06-13; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Palbociclib treatment
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib administration in breast cancer patients included in a compassionate use programme. Patients were treated according to the standard of care

SUMMARY:
In Spain, palbociclib was launched last November 1st, 2017. However, since February 2015 the on-going compassionate use programme of palbociclib has enabled drug access to patients with RH+/HER2- breast cancer previously treated with at least 4 treatment lines for advanced disease. During this period, approximately 400 patients have received treatment within this programme. Since this population of patients more pre-treated was not included in the studies for regulatory submission, the collection of efficacy and toxicity data in the clinical practice setting is of clinical interest.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RH+ y HER2- metastatic breast cancer having progressed to at least 4 previous standard treatment lines in the metastatic setting, and are not eligible to receive palbociclib in a clinical trial
2. Absolute neutrophil count ≥1,500/mm3 (1.5 x 109/L)
3. Platelet count ≥100,000/mm3 (100 x 109/L)
4. Haemoglobin ≥9 g/dL
5. Creatinine ≤1.5 x ULN or creatinine clearance ≥ 60 mL/min
6. Total bilirubin ≤1.5 x ULN (≤3.0 x ULN in case of Gilbert's disease)
7. AST and/or ALT ≤3 x ULN (≤5.0 x ULN in case of hepatic metastases)
8. Alkaline phosphatase ≤2.5 x ULN (≤5.0 x ULN in case of hepatic or bone metastases)

Exclusion Criteria:

1. Major surgery, chemotherapy, radiotherapy, treatment with an investigational drug or any other active anticancer therapy within two weeks of treatment initiation
2. Previous radiotherapy in ≥25% of bone marrow
3. QTc >480 msec, personal or family past history of short or long QT syndrome, Brugada's syndrome, or past history of QT interval prolongation, or tachycardia with Torsade de Pointes (TdP)
4. History of any of the following conditions within 6 months of treatment initiation: myocardial infarction, unstable angina, grade ≥2 arrhythmia (CTCAE version 4.0), atrial fibrillation, coronary or peripheral artery by-pass, symptomatic congestive heart failure, stroke, or pulmonary thromboembolism
5. Known hypersensitivity to palbociclib
6. Current or recent suicidal ideation or behaviour

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer included in a compassionate use programme
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Time to progression | through study completion, up to 9 months
  Number of days between the beginning of the treatment with palbociclib and the progression

SECONDARY OUTCOMES:
Number of adverse events | through study completion, up to 9 months
  Number of adverse events between the beginning of the treatment with palbociclib and the progression

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Moreno, Madrid, Spain